CLINICAL TRIAL: NCT03612713
Title: Influence of Medication on Functional Connectivity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2000020857; 1R21DA045969-01 (NIH); 1K01DA039299-01A1 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-08-02 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Prescription Drug Abuse (Not Dependent)
MeSH Terms: conditions — Substance-Related Disorders | interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxycodone Medication First (Active Comparator): one hour before fMRI scan participants will be given a single dose 15mg immediate release oxycodone
  Interventions: Drug: Oxycodone Medication First
- Placebo First (Placebo Comparator): one hour before fMRI scan participants will be given a single dose placebo.
  Interventions: Drug: Placebo First

INTERVENTIONS:
Drug: Oxycodone Medication First — Participants will be given 15mg oxycodone one hour before fMRI scan. After at least 1 week wash out participants will be given placebo one hour before fMRI scan.
  Other Names: Oxycodone
  Arms: Oxycodone Medication First
Drug: Placebo First — Participants will be given placebo one hour before fMRI scan. After at least 1 week wash out participants will be given 15mg oxycodone one hour before fMRI scan.
  Other Names: placebo
  Arms: Placebo First

SUMMARY:
This study will assess the effects of acute low-dose opioid administration on functional neuroimaging measures in healthy individuals

DETAILED DESCRIPTION:
This study will assess the effects of acute low-dose opioid administration on functional neuroimaging measures in healthy individuals (N=40, 20 male, 20 female). The objective of this research is to develop an understanding of factors that may influence individual variability on resting state functional connectivity in response to low-dose opioid administration with the longer term aim of understanding addictions vulnerability. Specifically, the proposed pilot research will explore the effects of single dose of oxycodone (15mg) on resting state functional connectivity and other common neuroimaging measures (e.g., diffusion MRI, structural MRI).

ELIGIBILITY:
Inclusion Criteria:

1. males or females, ages 18-30
2. for women of a child-bearing age, acceptable birth control methods or a negative pregnancy test prior to MRI scanning
3. ability to provide written, informed consent
4. eligibility and willingness to participate in fMRI scanning and to receive oxycodone
5. normal weight, as indicated by a body mass index (BMI) between 18.5 to 25

Exclusion Criteria:

1. current DSM-5 Axis I disorder
2. any psychotropic medication or medication known to interfere with metabolism of opioids
3. medical contraindication to participate in study activities (acute low-dose opioid admin) as determined by study physician
4. known family history (first-degree relative) of opioid-use disorder or alcohol-use disorder
5. not eligible for MRI scanning
6. positive drug screen
7. recent (past 6 months) medical or non-medical opioid-use
8. current or previous chronic pain disorder
9. significant lifetime use of prescription opioids (>7 days of consecutive medical use or nonmedical use on more than 5 occasions)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Yip, PhD, Principal Investigator — Yale University
Locations (1):
- Magnetic Resonance Research Center at The Anlyan Center Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxycodone Medication First | Placebo First
Started | 10 | 10
Completed | 7 | 8
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone Medication First | Placebo First | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.20 (2.82) | 24.40 (2.95) | 24.30 (2.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 6 | 9
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Connectivity Following Oxycodone Administration
Description: Functional connectivity is measured by functional magnetic resonance imagery (fMRI). Change in functional connectivity (a statistical relationship between two regions in the brain) between placebo and oxycodone fMRI scans will be assessed. Result is a transformed z-score. A score of 0 indicates no change. Higher scores indicate increased connectivity.
Time Frame: Change in functional connectivity from initial fMRI scan to follow-up MRI scan, up to 4 weeks.
Population: Positive and Negative connectivity within the ventral attention network
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Oxycodone Run: one hour before fMRI scan participants will be given a single dose 15mg immediate release oxycodone
- Placebo Run: one hour before fMRI scan participants will be given a placebo dose
Arm/Group | Oxycodone Run | Placebo Run
Number analyzed (Participants) | 12 | 12
z-score
  Positive network strength for connectivity within the ventral attention network | 2.66 (1.37) | 4.55 (2.46)
  Negative network strength for connectivity within the ventral attention network | .99 (.88) | 1.60 (.54)

ADVERSE EVENTS:
Time Frame: up to 4 weeks
Groups:
- Oxycodone Medication: one hour before fMRI scan participants will be given a single dose 15mg immediate release oxycodone
- Placebo: one hour before fMRI scan participants will be given a single dose placebo.
Arm/Group | Oxycodone Medication | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone Medication (N=20) | Placebo (N=20)
Nausea and vomiting (General disorders) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03612713/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03612713/ICF_001.pdf